CLINICAL TRIAL: NCT04257032
Title: Relative Bioavailability of Rosuvastatin (Part 1) and Dabigatran (Part 2) Given Alone and Together With BI 1323495 in Healthy Male Subjects (Open, Single-dose, Randomised, Two-period Crossover Design in Each Trial Part)
Brief Title: A Study in Healthy Men to Test the Influence of BI 1323495 on the Amount of the Medicines Rosuvastatin and Dabigatran in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1405-0015; 2019-004245-33 (EudraCT Number)
Record Dates: First submitted 2020-02-04; First posted 2020-02-05 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reference 1 (R1) (Experimental)
  Interventions: Drug: Rosuvastatin
- Test 1 (T1) (Experimental)
  Interventions: Drug: Rosuvastatin + BI 1323495
- Reference 2 (R2) (Experimental)
  Interventions: Drug: Dabigatran etexilate
- Test 2 (T2) (Experimental)
  Interventions: Drug: Dabigatran etexilate + BI 1323495

INTERVENTIONS:
Drug: Rosuvastatin — Tablet
  Arms: Reference 1 (R1)
Drug: Rosuvastatin + BI 1323495 — Tablets
  Arms: Test 1 (T1)
Drug: Dabigatran etexilate — Capsule
  Arms: Reference 2 (R2)
Drug: Dabigatran etexilate + BI 1323495 — Capsule and tablets
  Arms: Test 2 (T2)

SUMMARY:
The main objectives of this trial are to investigate the relative bioavailabilities of rosuvastatin (Reference 1, Part 1) and dabigatran (Reference 2, Part 2) given alone and together with BI 1323495 (Test 1, Test 2) following oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. BMI of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
5. Subjects genotyped as Uridine 5'-diphospho-Glucuronosyltransferase-2B17 (UGT2B17) extensive metabolisers, i.e. carrying at least one functional allele of UGT2B17 gene (*1/*1 or *1/*2)

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance (including positive or missing faecal occult blood test in Part 2)
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts
9. Chronic or relevant acute infections
10. History of relevant allergy or hypersensitivity (including allergy to the trial medications or their excipients)
11. Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial or compromise the subject's safety by participation in the trial (e. g. use of any drug that could reasonably inhibit platelet aggregation or coagulation, concomitant treatment with systemic cyclosporine, ketoconazole, itraconazole and dronedarone, use of fibrates or drugs that cause QT/QTc interval prolongation (QTc: QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTcB))
12. Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
13. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
14. Inability to refrain from smoking on specified trial days
15. Alcohol abuse (consumption of more than 24 g per day)
16. Drug abuse or positive drug screening
17. Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
18. Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
19. Inability to comply with the dietary regimen of the trial site
20. A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
21. A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
22. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
23. Male subjects with women of childbearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of administration of trial medication until 30 days thereafter. Sperm donation is not allowed from the time point of drug administration until 30 days thereafter.
24. Active clinically relevant bleeding or subjects who in the investigator's judgement are perceived as having an increased risk of bleeding, for example because of blood coagulation disorders, current or recent gastrointestinal ulceration, presence of malignant neoplasms, recent brain or spinal injury, recent brain/spinal/ophthalmic surgery, recent intracranial hemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms, major intraspinal or intracerebral vascular abnormalities
25. For Part 1 only: known myopathy, personal or family history of hereditary muscular disorders, or history of muscular toxicity with statins or fibrate; Asian ancestry; hypothyroidism
26. Subjects with any other condition that would preclude administration of rosuvastatin or dabigatran (i.e. contraindicated as per SmPC), such as active liver disease including elevations of serum transaminases exceeding 2 times the upper limit of normal, moderate or severe renal impairment (creatinine clearance < 60 ml/min based on estimated glomerular filtration rate (GFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula), prosthetic heart valves requiring anticoagulant treatment
27. During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open, single-dose, randomised, two-period, two way crossover design in each trial part to evaluate the relative bioavailability of rosuvastatin (Part 1) and dabigatran (Part 2) given alone and together with BI 1323495 in healthy male subjects.
Pre-assignment Details: All participants were entered/randomized for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all inclusion and none of the exclusion criteria. Subjects were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1323495 (T1): In part 1 (Reference (R1)- Test (T1)), on trial day 1 of period 1, a single oral dose of 1 film-coated tablet of 10 milligram (mg) rosuvastatin was administered with 240 milliliter (mL) of water after a standardised breakfast as reference treatment 1 (R1). Period 1 is followed by a washout period of at least 7 days. In part 1, on trial day 1 of period 2, a single oral dose of 1 film-coated tablet of 10 mg rosuvastatin was coadministered with a single oral dose of 6 film-coated tablets of 50 mg BI 1323495 (300 mg in total) with 240 mL of water after a standardised breakfast as test treatment 1 (T1).
- Part 1: Rosuvastatin + BI 1323495 (T1) / Rosuvastatin (R1): In part 1 (Test (T1)- Reference (R1)), on trial day 1 of period 1, a single oral dose of 1 film-coated tablet of 10 milligram (mg) rosuvastatin was coadministered with a single oral dose of 6 film-coated tablets of 50 mg BI 1323495 (300 mg in total) with 240 milliliter (mL) of water after a standardised breakfast as test treatment 1 (T1). Period 1 is followed by a washout period of at least 7 days. In part 1, on trial day 1 of period 2, a single oral dose of 1 film-coated tablet of 10 mg rosuvastatin was administered with 240 mL of water after a standardised breakfast as reference treatment 1 (R1).
- Part 2: Dabigatran (R2) / Dabigatran + BI 1323495 (T2): In part 2 (Reference (R2)- Test 2 (T2)), on trial day 1 of period 1, a single oral dose of 1 hard capsule of 75 milligram (mg) dabigatran etexilate was administered with 240 milliliter (mL) of water after a standardised breakfast as reference treatment 2 (R2). Period 1 is followed by a washout period of at least 7 days. In part 2, on trial day 1 of period 2, a single oral dose of 1 hard capsule of 75 mg dabigatran etexilate was coadministered with a single oral dose of 6 film-coated tablets of 50 mg BI 1323495 (300 mg in total) with 240 mL of water after a standardised breakfast as test treatment 2 (T2).
- Part 2: Dabigatran + BI 1323495 (T2) / Dabigatran (R2): In part 2 (Test 2 (T2) - Reference (R2)), on trial day 1 of period 1, a single oral dose of 1 hard capsule of 75 milligram (mg) dabigatran etexilate was coadministered with a single oral dose of 6 film-coated tablets of 50 mg BI 1323495 (300 mg in total) with 240 milliliter (mL) of water after a standardised breakfast as test treatment 2 (T2). Period 1 is followed by a washout period of at least 7 days. In part 2, on trial day 1 of period 2, a single oral dose of 1 hard capsule of 75 milligram (mg) dabigatran etexilate was administered with 240 milliliter (mL) of water after a standardised breakfast as reference treatment 2 (R2).
Period: Period 1 (+ Washout Period)
Arm/Group | Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1323495 (T1) | Part 1: Rosuvastatin + BI 1323495 (T1) / Rosuvastatin (R1) | Part 2: Dabigatran (R2) / Dabigatran + BI 1323495 (T2) | Part 2: Dabigatran + BI 1323495 (T2) / Dabigatran (R2)
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1323495 (T1) | Part 1: Rosuvastatin + BI 1323495 (T1) / Rosuvastatin (R1) | Part 2: Dabigatran (R2) / Dabigatran + BI 1323495 (T2) | Part 2: Dabigatran + BI 1323495 (T2) / Dabigatran (R2)
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1323495 (T1) | Part 1: Rosuvastatin + BI 1323495 (T1) / Rosuvastatin (R1) | Part 2: Dabigatran (R2) / Dabigatran + BI 1323495 (T2) | Part 2: Dabigatran + BI 1323495 (T2) / Dabigatran (R2) | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (10.3) | 44.3 (7.7) | 36.6 (10.3) | 35.7 (7.4) | 39.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 7 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 7 | 7 | 7 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve of the Analyte (Rosuvastatin) in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte (rosuvastatin) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Rosuvastatin (Reference 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration. Rosuvastatin + BI 1323495 (Test 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration.
Time Frame: Measured within 3 hours (h) before and up to 95h after drug administration. Detailed time frame is in description section.
Population: All subjects included in the Pharmacokinetic (PK) parameter analysis set (PKS) and with available data for this endpoint.
  PKS:All subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
  Rosuvastatin:AUC0-∞ only calculated for 12 subjects, due for 2 subjects concentrations at last sampling point were higher than at preceding time point.
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours * nanogramm / milliliter
Groups:
- Rosuvastatin (Part 1, Reference 1): In part 1 on study Day 1 of Period 1 or 2 a single oral dose of 1 film-coated tablet of 10 milligram (mg) rosuvastatin was administered with 240 milliliter (mL) of water after a standardised breakfast as reference 1 (R1).
- Rosuvastatin + BI 1323495 (Part 1, Test 1): In part 1 on study Day 1 of Period 1 or 2 a single oral dose of 1 film-coated tablet of 10 mg rosuvastatin was coadministered with a single oral dose of 6 film-coated tablets of 50 mg BI 1323495 (300 mg in total) with 240 mL of water after a standardised breakfast as test 1 (T1).
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1323495 (Part 1, Test 1)
Number analyzed (Participants) | 12 | 14
Hours * nanogramm / milliliter | 23.92 (NA) — (Adjusted) Geometric Standard Error = 1.13 | 25.20 (NA) — (Adjusted) Geometric Standard Error = 1.12
Statistical Analysis 1: Comparison: Rosuvastatin (Part 1, Reference 1) vs Rosuvastatin + BI 1323495 (Part 1, Test 1); Relative bioavailability; Test type: Other; ANOVA; ANOVA model on the logarithmic scale, considering the effects 'sequence', 'period' and 'treatment' as fixed and 'subjects within sequences' as random; Ratio of geometric means (T/R) % = 105.37, 90% CI 2-sided [97.94 to 113.35] — Intra-individual coefficient of variation (gCV %) = 9.9

2. Primary Outcome: Part 1: Maximum Measured Concentration of the Analyte (Rosuvastatin) in Plasma (Cmax)
Description: Maximum measured concentration of the analyte (rosuvastatin) in plasma (Cmax). Rosuvastatin (Reference 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration. Rosuvastatin + BI 1323495 (Test 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration.
Time Frame: as for outcome 1
Population: All subjects included in the Pharmacokinetic (PK) parameter analysis set (PKS) and with available data for this endpoint.
  PKS: All subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanogramm / milliliter
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1323495 (Part 1, Test 1)
Number analyzed (Participants) | 14 | 14
Nanogramm / milliliter | 2.20 (NA) — (Adjusted) Geometric Standard Error = 1.14 | 2.52 (NA) — (Adjusted) Geometric Standard Error = 1.14
Statistical Analysis 1: Comparison: Rosuvastatin (Part 1, Reference 1) vs Rosuvastatin + BI 1323495 (Part 1, Test 1); Relative bioavailability; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means (T/R) % = 114.50, 90% CI 2-sided [104.22 to 125.81] — Intra-individual coefficient of variation (gCV %) = 14.0

3. Primary Outcome: Part 2: Area Under the Concentration-time Curve of the Analyte (Dabigatran) in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte (dabigatran) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) Dabigatran (Reference 2) was measured within 3 hours (h) before drug administration and 30 minutes (min), 1h, 1h 30 min, 2h, 2h 30 min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 47h and 71h after drug administration. Dabigatran + BI 1323495 (Test 2) was measured within 3 hours (h) before drug administration and 30 minutes (min), 1h, 1h 30 min, 2h, 2h 30 min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 47h and 71h after drug administration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours * nanogramm / milliliter
Groups:
- Dabigatran (Part 2, Reference 2): In part 2 on study Day 1 of Period 1 or 2 a single oral dose of 1 hard capsule of 75 milligram (mg) dabigatran etexilate was administered with 240 milliliter (mL) of water after a standardised breakfast as reference 2 (R2).
- Dabigatran + BI 1323495 (Part 2, Test 2): In part 2 on study Day 1 of Period 1 or 2 a single oral dose of 1 hard capsule of 75 milligram (mg) dabigatran etexilate was coadministered with a single oral dose of 6 film-coated tablets of 50 mg BI 1323495 (300 mg in total) with 240 mL of water after a standardised breakfast as test 2 (T2).
Arm/Group | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1323495 (Part 2, Test 2)
Number analyzed (Participants) | 14 | 14
Hours * nanogramm / milliliter | 666.24 (NA) — (Adjusted) Geometric Standard Error = 1.08 | 720.76 (NA) — (Adjusted) Geometric Standard Error = 1.08
Statistical Analysis 1: Comparison: Dabigatran (Part 2, Reference 2) vs Dabigatran + BI 1323495 (Part 2, Test 2); Relative bioavailability; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means (T/R) % = 108.18, 90% CI 2-sided [100.26 to 116.73] — Intra-individual coefficient of variation (gCV %) = 11.3

4. Primary Outcome: Part 2: Maximum Measured Concentration of the Analyte (Dabigatran) in Plasma (Cmax)
Description: Maximum measured concentration of the analyte (dabigatran) in plasma (Cmax) Dabigatran (Reference 2) was measured within 3 hours (h) before drug administration and 30 minutes (min), 1h, 1h 30 min, 2h, 2h 30 min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 47h and 71h after drug administration. Dabigatran + BI 1323495 (Test 2) was measured within 3 hours (h) before drug administration and 30 minutes (min), 1h, 1h 30 min, 2h, 2h 30 min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 47h and 71h after drug administration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanogramm / milliliter
Arm/Group | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1323495 (Part 2, Test 2)
Number analyzed (Participants) | 14 | 14
Nanogramm / milliliter | 80.01 (NA) — (Adjusted) Geometric Standard Error = 1.08 | 87.12 (NA) — (Adjusted) Geometric Standard Error = 1.08
Statistical Analysis 1: Comparison: Dabigatran (Part 2, Reference 2) vs Dabigatran + BI 1323495 (Part 2, Test 2); Relative bioavailability; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means (T/R) % = 108.89, 90% CI 2-sided [99.84 to 118.76] — Intra-individual coefficient of variation (gCV %) = 12.9

5. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of the Analyte (Rosuvastatin) in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte (rosuvastatin) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  Rosuvastatin (Reference 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration. Rosuvastatin + BI 1323495 (Test 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 47h, 71h and 95h after drug administration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours * nanogramm / milliliter
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1323495 (Part 1, Test 1)
Number analyzed (Participants) | 14 | 14
Hours * nanogramm / milliliter | 21.50 (NA) — (Adjusted) Geometric Standard Error = 1.14 | 22.47 (NA) — (Adjusted) Geometric Standard Error = 1.14
Statistical Analysis 1: Comparison: Rosuvastatin (Part 1, Reference 1) vs Rosuvastatin + BI 1323495 (Part 1, Test 1); Relative bioavailability; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means (T/R) % = 104.52, 90% CI 2-sided [97.34 to 112.23] — Intra-individual coefficient of variation (gCV %) = 10.6

6. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of the Analyte (Dabigatran) in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte (dabigatran) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) Dabigatran (Reference 2) was measured within 3 hours (h) before drug administration and 30 minutes (min), 1h, 1h 30 min, 2h, 2h 30 min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 47h and 71h after drug administration. Dabigatran + BI 1323495 (Test 2) was measured within 3 hours (h) before drug administration and 30 minutes (min), 1h, 1h 30 min, 2h, 2h 30 min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 47h and 71h after drug administration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Hours * nanogramm / milliliter
Arm/Group | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1323495 (Part 2, Test 2)
Number analyzed (Participants) | 14 | 14
Hours * nanogramm / milliliter | 647.05 (NA) — (Adjusted) Geometric Standard Error = 1.08 | 701.55 (NA) — (Adjusted) Geometric Standard Error = 1.08
Statistical Analysis 1: Comparison: Dabigatran (Part 2, Reference 2) vs Dabigatran + BI 1323495 (Part 2, Test 2); Relative bioavailability; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means (T/R) % = 108.42, 90% CI 2-sided [100.37 to 117.12] — Intra-individual coefficient of variation (gCV %) = 11.5

ADVERSE EVENTS:
Time Frame: From the time of administration of test or reference treatment until administration time of next study drug dose or until 0:00 h on day 7 after time of administration, whatever occurs first, up to 7 days.
Description: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1323495 (Part 1, Test 1) | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1323495 (Part 2, Test 2)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/14 | 5/14 | 0/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin (Part 1, Reference 1) (N=14) | Rosuvastatin + BI 1323495 (Part 1, Test 1) (N=14) | Dabigatran (Part 2, Reference 2) (N=14) | Dabigatran + BI 1323495 (Part 2, Test 2) (N=14)
Fatigue (General disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT04257032/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04257032/SAP_001.pdf